CLINICAL TRIAL: NCT04236648
Title: Clinical and Radiographic Changes Following Minimally-invasive Non-surgical Therapy in Teeth With Unfavourable Prognosis: A Pilot Prospective Cohort Study
Brief Title: Minimally-invasive Non-surgical Treatment in Teeth With Unfavourable Prognosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perio-19-001
Record Dates: First submitted 2020-01-13; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally-invasive non-surgical therapy (MINST) (Other): Study treatment
  Interventions: Procedure: Minimally-invasive non-surgical therapy (MINST)

INTERVENTIONS:
Procedure: Minimally-invasive non-surgical therapy (MINST) — subgingival root debridement with a minimally-invasive approach using piezoelectric/ultrasonic instruments

SUMMARY:
This is a pilot prospective cohort study to assess the efficacy of minimally-invasive non-surgical periodontal therapy (MINST) for the treatment of teeth with unfavourable periodontal prognosis. 20 patients who have teeth with unfavourable periodontal prognosis (due to bone loss to the apex or furcation involvement grade II C) will receive minimally-invasive non-surgical treatment (MINST) and will be reassessed up to 12 months after treatment.

DETAILED DESCRIPTION:
Twenty patients with advanced periodontitis who have teeth with unfavourable periodontal prognosis (due to bone loss to the apex or furcation involvement grade II C) will be entered in this study, conducted at Guy's Hospital in London, UK. The study has a prospective cohort design, so following baseline assessment, all patients will receive minimally-invasive non-surgical treatment (MINST). A total of 10 visits are planned over a 12-13 months period including initial treatment (MINST) and follow-up appointments.

The primary outcomes are radiographic defect depth (for teeth with bone loss to the apex, n=10) and furcation involvement (for teeth with furcation involvement degree II C, n=10). Paired t-test will be used to detect significant changes between baseline and 12 months for the primary outcomes using the patient as unit of analysis. Additional outcomes will be probing pocket depths (PPD), clinical attachment level (CAL), levels of inflammatory markers and growth factors in gingival crevicular fluid (GCF) and saliva and bacterial detection in periodontal pockets

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Diagnosis of Periodontitis stage III or IV (grade A, B or C) (Tonetti et al. 2018)
* Presence of:
* N=10: Maxillary or mandibular molars with:

A. Furcation involvement degree II C based on Hamp et al. 1975 horizontal classification and Tarnow & Fletcher 1984 vertical classification (with concomitant furcation involvement (FI) not exceeding degree II on the other aspects of the same tooth) B. gingival recession ≤ 2mm on furcation site C. mobility maximum degree 2

* N=10: 'Teeth with bone loss to the apex' (also defined as 'hopeless' by Cortellini et al. 2011), defined as having:

A. radiographic bone loss to the apex or beyond the apex on at least one inter-dental aspect B. presence of severe attachment loss (>10 mm) at the same inter-proximal site/s and at least at one of either the buccal or lingual aspect (Cortellini et al. 2011) C. lack of function because of hypermobility, and/or lack of chewing strength, and/or pain, and/or recurrent periodontal infection/abscesses (Cortellini et al. 2011) D. positive response to vitality testing with electric pulp test (EPT) or previous endodontic treatment considered satisfactory, as judged by the examining clinician

- Willing to sign informed consent to take part in the study

Exclusion Criteria:

* Smoking (any current or in past 5 years)
* Medical history including diabetes or hepatic or renal disease, or other serious medical conditions or transmittable disease
* History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam
* Systemic antibiotic therapy during the 3 months preceding the baseline exam
* History of alcohol or drug abuse, vii) Self-reported pregnancy or lactation
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that according to the investigator may increase the risk associated with trial participation
* Periodontal treatment to the study site within the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic defect depth | baseline-12 months
  defect depth measured in radiographs in mm (as measured on standardised radiographs)
Furcation involvement | baseline-12 months
  furcation involvement measured clinically (as measured based on validated horizontal and vertical furcation involvement scales, by Hamp et al. 1975 and Tarnow 1984). Hamp et al. 1975 goes from 1 to 3 in increasing severity. Tarnow et al. score goes from A to C in increasing severity

SECONDARY OUTCOMES:
probing pocket depth | 0-12 months
  measure of gingival pocket depth (in mm with the use of University of North Carolina(UNC)-15 probe)
clinical attachment level | 0-12 months
  measure of pocket + gingival recession (in mm with use of UNC-15 probe)
patient-reported outcomes | 0-12 months
  Oral Health Impact Profile (OHIP)-14 questionnaire (standardised scale based on 14 questions). Each question can score from 0 to 4 in increasing severity (maximum total score can be 14x4= 56)
inflammatory response (in saliva and GCF) | 0-12 months
  measure of inflammatory cytokines (concentration in saliva and GCF), not restricted to some cytokines but explorative analyses of multiple cytokines by multiplex. The measure will be continuous, expressed for example in picograms/ml
subgingival microbes | 0-12 months
  analysis of presence of microbes subgingivally (metagenomic analysis)